CLINICAL TRIAL: NCT02422420
Title: Minnesota Medicaid Incentives to Prevent Chronic Disease
Acronym: MMIPCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnesota Department of Human Services (Other Government)
Collaborators: Minnesota Department of Health (Other Government); HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MinnesotaDHS; 1B1CMS330877-01-00 (Other: Centers for Medicare and Medicaid Services)
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-03

CONDITIONS: Prediabetic State
Keywords: Diabetes Prevention; Financial Incentives; Medicaid; Motivation
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Individual Incentive (Experimental): Participants receive a financial incentive every time they attend a class session and goal-based incentives for attending 75% of Core sessions, 75% of Post-Core sessions, separately achieving 5%, 7%, and 10% weight loss during the Core period (i.e. separate financial incentives for each goal reached at any point during the Core period), and 5%, 7%, or 10% weight loss by the end of Post-Core Session 8 (i.e., one financial incentive based on final weight loss).
  Interventions: Behavioral: Financial Incentives
- Group Incentive (Experimental): This arm receives the same routine attendance incentives as the Individual Incentive arm. Group goal-based incentives include 5% weight loss by an individual during the Core period and, separately, during the Post-Core period. Financial incentives are also received if the entire DPP group achieves 75% Core session attendance, 75% of Post-Core session attendance, 7% or 10% weight loss from baseline during the Core, and 7% or 10% weight loss from baseline at the end of the Post-Core period.
  Interventions: Behavioral: Financial Incentives
- Minimal Incentive (Other): Participants receive the full Diabetes Prevention Program (DPP), but receive a nominal $25 financial incentive for attendance only at the first DPP session and no other incentives for attendance or weight loss.
  Interventions: Behavioral: Financial Incentives

INTERVENTIONS:
Behavioral: Financial Incentives — Use of financial incentives to promote health behaviors.

SUMMARY:
The objective of this study is to test whether two different participant financial incentive structures are more effective and cost effective than minimal financial incentives in increasing weight loss among Minnesota Medicaid beneficiaries at high risk of developing diabetes. The incentives are tied to participation and weight loss in the evidence-based group-delivered YMCA diabetes prevention program (Y-DPP). The Investigators will conduct a group randomized trial that includes up to 150 Y-DPP classes of 10-15 participants per class for up to 1500 Medicaid beneficiaries participating in the Y-DPP classes. This approach, if successful, will (a) improve weight loss. diabetes risk, and improve cardiovascular risk among Medicaid beneficiaries at risk for developing diabetes and other chronic conditions, (b) demonstrate that prevention of chronic disease risk factors using patient incentives is cost-effective, and (c) provide a patient incentive model that can be widely used among Medicaid beneficiaries at risk for developing diabetes.

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled in Medical Assistance, PMAP, or MinnesotaCare (collectively referred to as Medicaid)
* 18-75 years of age
* body mass index ≥ 25 kg/m2 (≥ 22 kg/m2 for those of Asian descent)
* have prediabetes or a history of gestational diabetes mellitus (GDM)

Exclusion Criteria:

* diagnosis of diabetes
* pregnant at the time of enrollment
* planning gastric bypass surgery within the next 12 months
* diagnosed with Alzheimer's disease (ICD-9 331.0) or dementia (ICD-9 290.0 - 294.9)
* provider judgment regarding suitability for the study based on substance abuse, uncontrolled mental illness, or other conditions that may affect the participants health or ability to participate in the study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
DPP Attendance | 12 months
  Participation in DPP core and post-core sessions
Weight Change | 12 months
  Change in participants' weight

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Taylor, Principal Investigator — Minnesota Department of Health
Locations (1):
- Minnesota Department of Health, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Desai JR, Vazquez-Benitez G, Taylor G, Johnson S, Anderson J, Garrett JE, Gilmer T, Vue-Her H, Rinn S, Engel K, Schiff J, O'Connor PJ. The effects of financial incentives on diabetes prevention program attendance and weight loss among low-income patients: the We Can Prevent Diabetes cluster-randomized controlled trial. BMC Public Health. 2020 Oct 21;20(1):1587. doi: 10.1186/s12889-020-09683-5. PMID 33087083